CLINICAL TRIAL: NCT06805981
Title: Effects of Video-Based Cervical Posture and Breathing Exercises on Musculoskeletal System, Pain and Emotional Stress Levels in Young Adults
Brief Title: Effect of Telerehabilitation for Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Istanbul Gedik University (Other)
Responsible Party: Principal Investigator, ebrar atak, Asst. Prof., Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TeleRehabforYoungs
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2023-12

CONDITIONS: Young Adult Health
Keywords: Cervical posture exercises; Video-based exercise; Breathing exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- telerehabilitation group (Experimental): The study group received a total of 16 sessions of cervical posture exercises and breathing exercises, 30 minutes each session, twice a week for 8 weeks, using a video-based application together with a handout.
  Interventions: Other: telerehabilitation group
- Conventional rehabilitation group (Other): The control group was given a brochure containing cervical posture and breathing exercises. They were asked to do the exercises twice a week for 8 weeks, each session lasting 30 minutes, for a total of 16 sessions. Patient education was provided to the patients before rehabilitation.
  Interventions: Other: conventional rehabilitation group

INTERVENTIONS:
Other: telerehabilitation group — Asynchronous exercise videos were sent for follow-up for 8 weeks.
  Arms: telerehabilitation group
Other: conventional rehabilitation group — An exercise brochure with exercises to be followed for 8 weeks was given.
  Arms: Conventional rehabilitation group

SUMMARY:
It aims to examine the effects of video-based cervical posture and breathing exercises on the musculoskeletal system, pain and emotional stress levels in young adults. Control group (n: 15), study group (n: 15); It aims to examine the effects of video-based application support and breathing exercises and cervical posture exercises on the musculoskeletal health, which is important for individuals, pain affecting daily life and emotional stress levels, which we think have a great effect on social life, and to present them to the literature.

Primary Objective: To examine the effects of video-based cervical posture and breathing exercises on musculoskeletal health in young adults.

Secondary Objective: To examine the effects of video-based cervical posture and breathing exercises on pain in young adults.

Tertiary Objective: To examine the effects of video-based cervical posture and breathing exercises on emotional stress levels in young adults.

DETAILED DESCRIPTION:
The study will include 30 randomly selected individuals between the ages of 18 and 30 who were directed to the Istanbul Gedik University Physiotherapy and Rehabilitation Department laboratory.

The individuals included in the study will be divided into 2 groups as a control group and a study group of 15 people with simple randomization. Only a brochure will be given to the control group, and the brochure will be distributed and explained to the study group, and telerehabilitation will be applied.

The study will be carried out in the Istanbul Gedik University Physiotherapy and Rehabilitation Department laboratory.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 30 years old
* having enough technological equipment
* female - male gender
* volunteering to work

Exclusion Criteria:

* Those with vertigo
* those with frequent nausea
* those with severe dyspnea
* those with rib fractures

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Cornell Musculoskeletal System Questionnaire | Time duration of change eight week
  It evaluates the frequency of pain or discomfort in 11 different body parts during the day in the last week, the severity of this condition and its effect on work performance.
Cervical Posture Analysis | Time duration of change eight week
  Numerical data regarding general cervical posture (cervical lordosis, forward tilt of the head, etc.) will be obtained.
Neck Disability Index | Time duration of change eight week
  It is the most widely used assessment tool for measuring acute and chronic neck pain or disability due to neck injury.
Brief Pain Inventory | Time duration of change eight week
  It evaluates the severity of pain, the localization of pain, medical treatments for pain, and the effect of pain on daily functions, and asks how much pain has decreased in the last 24 hours or the last week.

CONTACTS AND LOCATIONS:
Overall Officials: Amine Ataç, Asst. Prof., Principal Investigator — amineatac@gmail.com
Locations (1):
- Ebrar Atak, Yalova, Türkiye/Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be evaluated if the researchers are contacted via their e-mail addresses.

REFERENCES:
- [Background] Bourne S, DeVos R, North M, Chauhan A, Green B, Brown T, Cornelius V, Wilkinson T. Online versus face-to-face pulmonary rehabilitation for patients with chronic obstructive pulmonary disease: randomised controlled trial. BMJ Open. 2017 Jul 17;7(7):e014580. doi: 10.1136/bmjopen-2016-014580. PMID 28716786